CLINICAL TRIAL: NCT04504747
Title: Real Time Molecular Analysis of Breast Cancer Receiving Neo-adjuvant Chemotherapy: Identification of Preclinical Models Predictive for Therapeutic Resistance
Brief Title: Real Time Molecular Analysis of Breast Cancer Receiving Neo-adjuvant Chemotherapy
Acronym: NEO-R
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: NEO-R-IPC 2019-041
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Tumor Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bllod and tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- RH+: Prospective blood and biopsie analyses
  Interventions: Other: molecular analysis of blood and tumor
- HER2+: Prospective blood and biopsie analyses
  Interventions: Other: molecular analysis of blood and tumor
- TN: Prospective blood and biopsie analyses
  Interventions: Other: molecular analysis of blood and tumor

INTERVENTIONS:
Other: molecular analysis of blood and tumor — RNAseq, DNAseq, CTCs

SUMMARY:
The present project aims at identifying robust candidates for drug resistance in BC patients eligible for NAC. Its originality lies upon the combination of three different and complementary prospective approaches: from the molecular analyses of biopsies sampled before and after NAC, from in vitro BC Patient-Derived Organoids (PDO) mimicking patient's response to NAC, and from Circulating Tumor Cells (CTCs) isolated before/during/after NAC.

DETAILED DESCRIPTION:
Breast cancer (BC) is a major public health problem in France, with an increasing incidence, estimated at ~60,000 new cases in 2017 and 12,000 deaths. Despite survival improvement in the recent years, resistance to chemotherapy (CT) remains a paramount challenge in BC: the molecular mechanisms remain poorly known and the current interventions are inadequate to target chemoresistance. Neo-adjuvant chimiotherapy (NAC) is now used increasingly in women with operable but aggressive BC such as triple-negative (TN) or HER2+ tumor (Pusztai et al, Lancet Oncol 2019). It provides at least three advantages: i) tumor debulking authorizing conservative surgery, ii) tailoring of adjuvant systemic therapy according to the pathological response, with delivery of capecitabine in TN patients (Masuda N. et al, N Engl J Med. 2017) and T-DM1 in HER2+ patients (von Minckwitz G et al., N Engl J Med. 2019) in the absence of pathological complete response (pCR), and iii) providing resources for investigating the molecular mechanisms of chemoresistance. The current standard NAC regimen is based on a sequential association of anthracycline and taxane (and trastuzumab if HER2+) (Huober & von Minckwitz, Breast Care 2011), and the achievement of pCR, defined as the absence of residual invasive cancer on pathological evaluation of the operative specimen (resected breast specimen and sampled ipsilateral lymph nodes (i.e., ypT0/Tis ypN0 in the AJCC staging system), is a good-prognosis feature; the patients without pCR being at high relapse risk (≈50% of the TN and HER2+ subtypes).

The major bottleneck in improving treatment efficiency for these patients is the identification of candidates effectively involved in the resistance to NAC, their validation in relevant and predictive models, and their detection from surrogate markers. Of course, the search for molecular alterations differentially represented in the pre-NAC samples between the resistant (no pCR) versus sensitive (pCR) patients, or between the paired post- versus pre-NAC samples may reveal candidates involved in resistance ("innate" and "acquired stable" respectively), but ignores the alterations that occur during the NAC that may be reversible ("acquired reversible") and not identified in the resected specimen (Echeverria GV, Sci Transl Med 2019), but only identifiable by analysis of serial samples during NAC regimen, difficult and traumatic in clinical practice.

The present project aims at identifying robust candidates for drug resistance in BC patients eligible for NAC. Its originality lies upon the combination of three different and complementary prospective approaches: from the molecular analyses of biopsies sampled before and after NAC, from in vitro BC Patient-Derived Organoids (PDO) mimicking patient's response to NAC, and from Circulating Tumor Cells (CTCs) isolated before/during/after NAC. This project will combine the most advanced technologies (RNA and DNA-sequencing from small amount of biologic material, rare subsets/single-cell isolation, and multi-omics analyses) with innovative models (drug testing on breast PDO, identification of reversible drug-induced changes) and clever combination of robust markers involved in drug resistance that have all been established and are running in the laboratory (cf Part B). The last two points have only recently become feasible thanks to two recent technological advances: breast cancer PDO cultures (Sachs N, et al. Cell. 2018) and CTCs isolation and characterization (Gkountela S, et al. Cell. 2019). Briefly, the investigators will use serial tumor biopsies and blood samples from a cohort of BC patients treated with NAC (Figure 1). Tumor biopsies will be collected before and after NAC. They will be analyzed by RNA-seq and targeted-NGS (exome) approaches to capture the differences resulting from NAC in patients with different pathological response. They will also be used to generate BC PDO models. The PDO models predictive for NAC response will be exploited as relevant models to investigate NAC resistance. Specifically, investigators will use these models to look at in vitro "acquired reversible" drug-induced resistance mechanisms (i.e only detectable during the drug exposure). Blood samples will be collected before, during, and after NAC to analyze CTCs, and aim at identifying "acquired reversible" drug-induced resistance mechanisms ex vivo, which the investigators might fail to detect with the before/after NAC samples only.

To our knowledge, this is the first time that these three innovative approaches will be used together to investigate in depth the topic of "resistance" in patients receiving NAC. The strength of this combination is to anticipate different - not mutually exclusive - situations that might occur ("innate", "acquired stable" and/or "reversible" drug-induced resistance). Each approach will provide original, precise and specific information that will contribute to build a more complete answer to this question than the scattered and incomplete data currently available in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Woman over 18
2. Signed consent to participate
3. Invasive mammary adenocarcinoma proven histologically and / or cytologically
4. Indication of CNA retention by the referring clinical team.
5. No contraindication to CNA.
6. Selected indication of the post-CNA surgery sequence, then radiotherapy
7. Performance index ≤ 1 (WHO).
8. Affiliation to a social security scheme, or beneficiary of such a scheme

Exclusion Criteria:

1. Planned therapeutic sequence: CNA, followed by neoadjuvant radiotherapy (HIST-RIC clinical trial for example) before surgery
2. Metastatic disease at diagnosis
3. Patient relapsed from breast cancer precede
4. Other malignant disease in the previous 3 years, with the exception of cervical carcinoma in situ or skin basal cell carcinoma and any other cancerous pathology considered to have been properly treated and at low risk of relapse.
5. Woman pregnant or likely to be (without effective contraception) or breastfeeding
6. Person in an emergency situation, adult person subject to a legal protection measure (adult under guardianship, guardianship or legal protection), or unable to express consent.
7. Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brest cancer females with a non metastatic cancer
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Identify robust candidates - "innate, "acquired stable" and/or reversible" | 5 years
  comparison of pre and/or post NAC molecular profiles in tumors, PDO models and CTCs - will be targeted with a drug in relevant models

SECONDARY OUTCOMES:
public repertoire of whole transcriptome and targeted-NGS | 5 years
  NAC" database will be constructed from well documented RNAseq and targeted-NGS profiles established from serial HER2+ and TN tumors before/after NAC treatment
Identify molecular signatures associated with response to NAC | 5 years
  Comparison of serial molecular profiles
Establish PDO samples exposed to NAC | 5 years
  Percentage of PDO exposed to NAC that will parallel the patient's clinical response to NAC
Evaluation of CTCs features | 5 years
  phenotype, RNA-seq-based transcriptome

CONTACTS AND LOCATIONS:
Overall Officials: François BERTUCCI, Pr, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No